CLINICAL TRIAL: NCT06802731
Title: A Multicenter Study on the Application of LivQ-box® Parameters in the Diagnosis of Liver Inflammation in Patients with Non-alcoholic Fatty Liver Disease
Brief Title: LivQ-box® Parameters in the Diagnosis of Liver Inflammation
Status: Recruiting | Type: Observational
Sponsor: Wuxi Hisky Medical Technology Co Ltd (Industry)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HSKE-LI001
Record Dates: First submitted 2025-01-13; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Liver Inflammation; Fatty Liver Disease
MeSH Terms: conditions — Hepatitis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the correlation between LivQ-box® parameters carried by iLivTouch and liver inflammation in patients with NAFLD, as well as the diagnostic value of liver inflammation of different severity levels.

DETAILED DESCRIPTION:
This study is a multi-center study that retrospectively analyzed and prospectively included 240 NAFLD patients in total who met the inclusion criteria. The laboratory, iLivTouch, and liver biopsy results were collected to evaluate the correlation between LivQ-box® parameters carried by iLivTouch and liver inflammation in patients with NAFLD, as well as the diagnostic value of liver inflammation of different severity levels. In the end, cut-off values for different stages of inflammation were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with NAFLD according to The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases;
* Age over 18 years old, gender not limited;
* Not combined with liver diseases (such as viral hepatitis, drug-induced liver injury, autoimmune liver disease);
* Perform iLivTouch examination within ± 14 days of liver pathology examination;
* No history of excessive alcohol consumption (converted to ethanol:<140g/week for males,<70g/week for females);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NAFLD according to The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the correlation and diagnostic performance of LivQ-box and cut-off values for different inflammation stages in NAFLD patients based on iLivTouch. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital (BTCH) affiliated to Tsinghua University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Negro F. Natural history of NASH and HCC. Liver Int. 2020 Feb;40 Suppl 1:72-76. doi: 10.1111/liv.14362. PMID 32077608
- [Background] Zhou J, Zhou F, Wang W, Zhang XJ, Ji YX, Zhang P, She ZG, Zhu L, Cai J, Li H. Epidemiological Features of NAFLD From 1999 to 2018 in China. Hepatology. 2020 May;71(5):1851-1864. doi: 10.1002/hep.31150. PMID 32012320
- [Background] Man S, Deng Y, Ma Y, Fu J, Bao H, Yu C, Lv J, Liu H, Wang B, Li L. Prevalence of Liver Steatosis and Fibrosis in the General Population and Various High-Risk Populations: A Nationwide Study With 5.7 Million Adults in China. Gastroenterology. 2023 Oct;165(4):1025-1040. doi: 10.1053/j.gastro.2023.05.053. Epub 2023 Jun 26. PMID 37380136
- [Background] Oda K, Uto H, Mawatari S, Ido A. Clinical features of hepatocellular carcinoma associated with nonalcoholic fatty liver disease: a review of human studies. Clin J Gastroenterol. 2015 Feb;8(1):1-9. doi: 10.1007/s12328-014-0548-5. Epub 2015 Jan 10. PMID 25575848
- [Background] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287
- [Background] Alexander M, Loomis AK, van der Lei J, Duarte-Salles T, Prieto-Alhambra D, Ansell D, Pasqua A, Lapi F, Rijnbeek P, Mosseveld M, Waterworth DM, Kendrick S, Sattar N, Alazawi W. Risks and clinical predictors of cirrhosis and hepatocellular carcinoma diagnoses in adults with diagnosed NAFLD: real-world study of 18 million patients in four European cohorts. BMC Med. 2019 May 20;17(1):95. doi: 10.1186/s12916-019-1321-x. PMID 31104631
- [Background] Estes C, Anstee QM, Arias-Loste MT, Bantel H, Bellentani S, Caballeria J, Colombo M, Craxi A, Crespo J, Day CP, Eguchi Y, Geier A, Kondili LA, Kroy DC, Lazarus JV, Loomba R, Manns MP, Marchesini G, Nakajima A, Negro F, Petta S, Ratziu V, Romero-Gomez M, Sanyal A, Schattenberg JM, Tacke F, Tanaka J, Trautwein C, Wei L, Zeuzem S, Razavi H. Modeling NAFLD disease burden in China, France, Germany, Italy, Japan, Spain, United Kingdom, and United States for the period 2016-2030. J Hepatol. 2018 Oct;69(4):896-904. doi: 10.1016/j.jhep.2018.05.036. Epub 2018 Jun 8. PMID 29886156
- [Background] Wong VW, Wong GL, Tsang SW, Hui AY, Chan AW, Choi PC, Chim AM, Chu S, Chan FK, Sung JJ, Chan HL. Metabolic and histological features of non-alcoholic fatty liver disease patients with different serum alanine aminotransferase levels. Aliment Pharmacol Ther. 2009 Feb 15;29(4):387-96. doi: 10.1111/j.1365-2036.2008.03896.x. Epub 2008 Nov 17. PMID 19035982
- [Background] Harris R, Harman DJ, Card TR, Aithal GP, Guha IN. Prevalence of clinically significant liver disease within the general population, as defined by non-invasive markers of liver fibrosis: a systematic review. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):288-297. doi: 10.1016/S2468-1253(16)30205-9. Epub 2017 Feb 1. PMID 28404158
- [Background] Gao F, He Q, Li G, Huang OY, Tang LJ, Wang XD, Targher G, Byrne CD, Luo JW, Zheng MH. A novel quantitative ultrasound technique for identifying non-alcoholic steatohepatitis. Liver Int. 2022 Jan;42(1):80-91. doi: 10.1111/liv.15064. Epub 2021 Sep 30. PMID 34564946